CLINICAL TRIAL: NCT03260699
Title: To Determine the Economic and Functional Impact of Peri-Operative Extension Assist Pneumatic Bracing for Primary Total Knee Arthroplasty (TKA) Non-Inferiority Trial
Brief Title: Economic and Functional Impact of Peri-Operative Bracing for Primary Total Knee Arthroplasty (TKA)
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated per Ongoing Care Solutions, Inc.
Sponsor: The Cleveland Clinic (Other)
Responsible Party: Principal Investigator, Carlos Higuera-Rueda, Staff Surgeon, The Cleveland Clinic
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SHB-OCSI007
Record Dates: First submitted 2017-07-10; First posted 2017-08-24 (Actual); Results first posted 2019-08-14 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-09

CONDITIONS: Arthropathy of Knee

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Control group (No Intervention): Subjects will receive two out-patient physical therapy (PT) visits per week for 2 weeks, followed by additional PT visits at clinician's discretion after TKA.
- Bracing group (Experimental): Subjects will be fitted with the Ongoing Care Solutions, Inc (OCSI) Rehabilitator brace prior to surgery. This brace will be worn for 6 weeks before surgery. The brace will be worn again after surgery ~10 days after surgery or when staples are removed until the end of the study. Participants will also have two PT visits per week for 2 weeks, followed by additional PT visits at clinician's discretion.
  Interventions: Device: OCSI Rehabilitator brace

INTERVENTIONS:
Device: OCSI Rehabilitator brace — Guardian Brace features the innovative Rehabilitator™ line of gait correcting, leg strengthening braces. Rehabilitator™ Knee Braces are clinically proven to reduce UNBRACED pain, strengthen the affected leg, and significantly improve function after only 90 days of brace wear.
  Arms: Bracing group

SUMMARY:
While bracing has been shown to be beneficial for patients with osteoarthritis (OA) in terms of function and strength, whether these unloader braces are also similarly beneficial after total knee arthroplasty (TKA) surgery needs to be examined. Therefore the investigators questioned whether wearing a brace that has previously been shown to increase strength and function in OA patients can also increase strength and function in patients after TKA.

ELIGIBILITY:
Inclusion Criteria:

Age: 50 years or older

Exclusion Criteria:

* BMI > 40
* Radiographic deformity of greater than 10 degrees

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2017-10-05 (Actual); Primary Completion 2018-01-01 (Actual); Study Completion 2018-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Spindler Kurt, MD, Study Chair — Department Chair
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bracing Group: Subjects will be fitted with the Ongoing Care Solutions, Inc (OCSI) Rehabilitator brace prior to surgery. This brace will be worn for 6 weeks before surgery. The brace will be worn again after surgery ~10 days after surgery or when staples are removed until the end of the study. Participants will also have two PT visits per week for 2 weeks, followed by additional PT visits at clinician's discretion.
  OCSI Rehabilitator brace: Guardian Brace features the new Rehabilitator™ line of gait correcting, leg strengthening braces. It is hypothesized that this brace may help reduce pain and improve knee function.
Period: Overall Study
Arm/Group | Control Group | Bracing Group
Started | 5 | 4
Completed | 5 | 2
Not Completed | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Bracing Group | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 4 | 1 | 5
  >=65 years | 1 | 3 | 4
Age, Continuous [Mean (Full Range); unit: years] | 64.2 [60 to 71] | 67.7 [63 to 73] | 65 [60 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 3 | 3
  Male | 5 | 1 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 5 | 1 | 6
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 9
Body-mass Index [Mean (Full Range); unit: kg/m^2] | 34.3 [28.7 to 39.75] | 26.9 [21.41 to 30.56] | 31 [21.41 to 39.75]

OUTCOME MEASURES:

1. Primary Outcome: Number of Physical Therapy Visits
Description: Investigators will monitor the total number of physical therapy visits that was necessary to return to normal function between the control and bracing group and how it relates to overall cost.
Time Frame: Total number of visits from date of surgery to 12 weeks after surgery
Measure: Mean (Full Range); unit: visit
Arm/Group | Control Group | Bracing Group
Number analyzed (Participants) | 5 | 2
visit | 14 [6 to 22] | 4 [2 to 5]

2. Secondary Outcome: Visual Analog Scale (VAS) for Pain (0-10 Scale)
Description: Visual Analog Scale is a a pain scale assessment instrument that has been widely used to allow adult patients to report their pain level in musculoskeletal research studies. It is a continuous scale comprised of a horizontal line, 10 centimeters (100 mm) in length, anchored by 2 two ends representing the extremes of measurements with 0 point representing no pain and 10 representing the worst pain a patient may have had. Therefore, starting from zero point, increasing numbers demonstrate worse pain. Patient can pick a point on the scale that they believe represent their pain level at a given moment.
Time Frame: Change from baseline to 12 weeks after surgery
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control Group | Bracing Group
Number analyzed (Participants) | 5 | 2
units on a scale | 3 [2 to 4] | 2 [1 to 3]

3. Secondary Outcome: Timed up and go Test (Timed Measurement)
Description: Used to assess a person's mobility and balance. It is measured in time units (seconds or minutes) using a stopwatch by a study personnel. To perform, the patient sits back in a standard arm chair and a line 3 meters, or 10 feet away on the floor is identified. At the investigator mark, the stopwatch is started and the patient is asked to stand up from chair, walk to the end of the line and come back to his chair at normal pace. The results is the time in seconds needed for the patient to perform the test (getting up from chair and coming back to it as timed by the investigator's stopwatch)
Time Frame: Change from baseline to 12 weeks after surgery
Measure: Mean (Full Range); unit: Seconds
Arm/Group | Control Group | Bracing Group
Number analyzed (Participants) | 5 | 2
Seconds | 4 [2 to 6] | 10 [6 to 14]

4. Secondary Outcome: Timed Stair Climb (Timed Measurement Over Fixed Distance)
Description: Used to assess a person's mobility and balance
Time Frame: Change from baseline to 12 weeks after surgery
Measure: Mean (Full Range); unit: seconds
Arm/Group | Control Group | Bracing Group
Number analyzed (Participants) | 5 | 2
seconds | 10 [8 to 12] | 17 [15 to 19]

5. Secondary Outcome: One-leg Stance Time (Timed Measurement)
Description: Used to assess a person's balance. Performed with eyes open and arms on hips. The patient is asked to stand unassisted on one leg and is timed in seconds (using stopwatch) from the time one foot is flexed off the floor to the time when it touches the ground or the standing leg or an arm leaves the hips.
Time Frame: Change from baseline to 12 weeks after surgery
Measure: Mean (Full Range); unit: seconds
Arm/Group | Control Group | Bracing Group
Number analyzed (Participants) | 5 | 2
seconds | 21 [13 to 29] | 32 [30 to 34]

6. Secondary Outcome: 6 Minute Walk Test (Distance Measurement)
Description: Used to assess a person's endurance and aerobic capacity. The score of the test is distance a patient walks in 6 minutes. Longer distances walked by the patient in 6 minutes correlates with better performance. Distance is measured using distance measuring wheel.
Time Frame: Change from baseline to 12 weeks after surgery
Measure: Mean (Full Range); unit: meters
Arm/Group | Control Group | Bracing Group
Number analyzed (Participants) | 5 | 2
meters | 68 [60 to 79] | 89 [80 to 89]

7. Secondary Outcome: Knee Society Score Questionnaire
Description: Clinical outcome questionnaire developed by the consensus of the Knee Society. It comprises, a "Knee score" and a "Functional score." The Knee score assesses pain, stability, and range of motion. A maximum score of 100 is achieved by a painless, well-aligned knee with 125° range of motion, with neither anteroposterior nor mediolateral instability. Deductions are made for flexion contracture, extension lag, and malalignment. The Functional score assesses walking distance and stair climbing. A maximum score of 100 is assigned to individuals who can walk unlimited distances and can climb up and down stairs normally. Deductions are made for use of a walking stick or crutches. Therefore, higher scores correlate with better function and outcome.
Time Frame: Change from baseline to 12 weeks after surgery
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control Group | Bracing Group
Number analyzed (Participants) | 5 | 2
units on a scale | 29 [23 to 36] | 33 [29 to 37]

8. Secondary Outcome: Knee Injury and Osteoarthritis Outcome Score Jr. (KOOS Jr.) Questionnaires
Description: Clinical outcome questionnaire that measure joint-specific pain and physical function. It has seven questions that focus on three categories: joint pain, stiffness, and function, in daily living. Raw scores are added up (range 0-28) and converted to an interval score (0-100) using an interval table. The interval score represents a patients total joint disability where 0 corresponds to total joint disability and 100 perfect joint health.
Time Frame: Change from baseline to 12 weeks after surgery
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control Group | Bracing Group
Number analyzed (Participants) | 5 | 2
units on a scale | 35 [28 to 42] | 41 [39 to 43]

9. Secondary Outcome: Hospital for Special Surgery (HSS) Score (0-100 Scale)
Description: Clinical outcome assessment tool. It is based on a total of 100 points. The score is divided into seven categories, which include pain, function, range of motion, muscle strength, flexion deformity, instability, and subtractions. The knee is initially given a score of 0, and additions or subtractions are made according to specific criteria. The higher the score, the better the outcome. Approximately 50% of the score is based on a patient interview and the remaining on physical exam.
Time Frame: Change from baseline to 12 weeks after surgery
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Control Group | Bracing Group
Number analyzed (Participants) | 5 | 2
units on a scale | 21 [15 to 27] | 21 [17 to 25]

10. Secondary Outcome: Type of Pain Medication Used
Description: Investigators will monitor the medical record for types of pain medications used.
Time Frame: Change from baseline to 12 weeks after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Bracing Group
Number analyzed (Participants) | 5 | 2
Participants
  Patients who used opioids | 5 | 2
  Patients who did not use opioid medications | 0 | 0

11. Secondary Outcome: Amount of Pain Medication Used
Description: Investigators will monitor the medical record for the amount of pain medication used
Time Frame: Change from baseline to 12 weeks after surgery
Measure: Mean (Standard Deviation); unit: morphine equivalents/day
Arm/Group | Control Group | Bracing Group
Number analyzed (Participants) | 5 | 2
morphine equivalents/day | 30 (8) | 45 (8)

ADVERSE EVENTS:
Time Frame: 9 months postoperative for each patient
Description: Definitions are similar to clinicaltrials.gov. Systmatic assessment was performed for patients with follow-up visit and at the 9 months point for each by chart review. The adverse events were then recorded for the cohort.
Arm/Group | Control Group | Bracing Group
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/2
Other Adverse Events (participants affected / at risk) | 2/5 | 1/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=5) | Bracing Group (N=2)
Transient right sided numbness (Nervous system disorders) | 0 (0) | 1 (3)
Knee stiffness (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Shortness of breath (Cardiac disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-05): https://cdn.clinicaltrials.gov/large-docs/99/NCT03260699/Prot_SAP_000.pdf